CLINICAL TRIAL: NCT01870310
Title: Long Term Study on the Possible Beneficial Effects of Catheterised Renal Denervation in Patients With Heart Failure and Left Ventricular Systolic Dysfunction Who Are Already on Standard Medical Therapy.
Brief Title: Renal Denervation in Patients With Heart Failure and Severe Left Ventricular Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, doc. MUDr. Miloš Táborský, CSc., FESC, MBA, Head of Department of First Clinic of Internal Medicine - Cardiology, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLOMOUC 1
Record Dates: First submitted 2013-05-25; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure
Keywords: Heart failure; Renal denervation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard medical therapy (No Intervention)
- Renal denervation + standard medical therapy (Experimental): Patients in this arm will undergo catheterised renal denervation in addition to having optimization of medical therapy for heart failure.
  Interventions: Procedure: Catheterised renal denervation

INTERVENTIONS:
Procedure: Catheterised renal denervation
  Other Names: Symplicity, Ardian / Medtronic, USA
  Arms: Renal denervation + standard medical therapy

SUMMARY:
It is a randomized prospective controlled study evaluating the effect of transcatheter renal denervation on the clinical status of patients with chronic heart failure and its safety procedures. The working hypothesis of the study is that by performing transcatheter renal denervation in patients with chronic heart failure and severe left ventricular systolic dysfunction there will a resultant reduction in the renal sympathetic activation which in turn will reduce the number of hospitalizations and deaths from heart failure.

DETAILED DESCRIPTION:
Chronic heart failure in the European countries occurs in 2-3% of the population with a significant increase in the higher age groups (1). Improved treatment of acute conditions (especially myocardial infarction) has resulted in more patients entering into the category of chronic heart failure. Chronic heart failure has a poor prognosis. Diagnosis and treatment are challenging both medically and economically. Half of the patients with systolic heart failure die within 4 years and more than 50% of patients with severe heart failure (NYHA functional class of IV) die within one year (1). The current treatments for heart failure are not only aimed at influencing the symptoms, but also preventing the progression of heart failure to reduce mortality.

Heart failure leads to the activation of compensatory mechanisms designed to restore adequate cardiac output. These mechanisms are initially beneficial, but their long-term activation leads to further progression of the pathological process and deterioration of cardiac function. One of the basic pathophysiological processes in heart failure is excessive activation of the sympathetic nervous system. This causes increased levels of circulating catecholamines which is proportional to the severity of the disease that is patients with the highest levels of norepinephrine have the worst prognosis. Beta-blocker therapy which is designed to inhibit activity of sympathetic nervous system causes milder symptoms of heart failure in patients by modifying disturbed hemodynamics and ultimately the clinical status. In recent years, the therapeutic efficacy of beta-blockers in chronic heart failure has been verified in a number of controlled clinical trials (2-5). These studies have confirmed that long-term treatment with beta-blocker therapy alleviates the symptoms of heart failure, improves the clinical condition of the patients and reduces mortality like ACE inhibitors.

High activity of renal sympathetic nerves in patients with chronic heart failure is an early predictor of increased mortality (6). The main pathophysiological basis of this finding is probably excessive sodium retention due to direct activation of sympathetic fibers innervating renal tubules (7). Recent experimental work on animals have shown that surgical renal denervation inhibits an increase in renal vascular resistance, prevents a decrease in renal blood flow (8), and also prevents changes in expression of angiotensin receptors in the kidney (8).

Surgical sympathectomy began to be used for the treatment of severe and malignant hypertension more than 50 years ago. But this was a rather complicated procedure, which was accompanied by a number of adverse effects (orthostatic hypotension and tachycardia, shortness of breath, bowel and sexual disorders]. Moreover it required a long hospitalization of 2-4 weeks and then required a recovery period of 1-2 months. However this intervention led to a rapid decrease in pressure and a higher survival rate after surgery in a large observational study(9).

In recent years a method has been developed in which destruction of renal sympathetic nerves that are present in the adventitia of renal arterial walls is done by catheterization (10). This procedure uses a catheter with a radiofrequency ablator at its tip (Symplicity, Ardian / Medtronic, USA), which is introduced through the femoral artery and then progressively introduced into the renal arteries. A randomized study has demonstrated that this procedure has a high degree of safety for the patients and a high rate of efficacy as well. In patients with resistant hypertension treated with transcatheter renal denervation there was a significant drop in blood pressure of 33/11 mmHg (p < 0.0001) that occurred after 6 months compared to a control group receiving unmodified pharmacological treatment (11).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with chronic heart failure, ischemic and non-ischemic etiology.
* NYHA (New York Heart Association) class II-IV.
* LVEF (Left Ventricular Ejection Fraction) ≤ 35%.
* Patients treated with maximum tolerated doses of standard pharmacotherapy for heart failure, who were stable for at least four weeks without acute decompensated heart failure.
* Prior to enrollment, patients must give informed consent.

Exclusion Criteria:

* Patients with history of acute coronary syndrome or stroke within the last 6 months.
* Significant valvular defects and/or planned cardiac surgery.
* Systolic blood pressure <110 mmHg.
* Advanced renal insufficiency (estimated GFR (Glomerular Filtration Rate) according to MDRD <30 ml/min/1.73 square meters).
* Unsuitable anatomy of renal arteries (presence of significant renal stenosis, renal artery narrower than 4 mm).
* Patients who underwent renal angioplasty or stent placement into the renal artery in the past.
* Severe coagulation disorders.
* Pregnancy or lactation.
* Refusal of the patient.
* Other diseases limiting prognosis of the patient to less than 2 years.
* Other reasons which in the opinion of the attending physician would preclude the individual from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-09 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum NT-proBNP at 6 months and 1 year from baseline in both groups. | 6 months and 1 year
  The level of NT-proBNP (N-terminal prohormone of Brain Natriuretic Peptide) is a reliable indicator of the severity of heart failure. Lowering levels will indicate improvement in the heart function.

SECONDARY OUTCOMES:
Reduction in the number of hospitalizations and/or deaths due to cardiovascular causes. | 1 year to 4 years

OTHER OUTCOMES:
Significant Renal impairment and symptomatic hypotension. | 6 months to 1 year
  Increase in serum creatinine of 2 times the baseline or decrease in estimated glomerular filtration according to MDRD (Modification of Diet in Renal Disease) by more than 50% from baseline will be used to assess renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Miloš Táborský, doc., MUDr., CSc., FESC, MBA, Principal Investigator — Head of Department of First Clinic of Internal Medicine - Cardiology, University Hospital, Olomouc.
Locations (1):
- University Hospital, Olomouc, Olomouc, Olomouc, Czechia

REFERENCES:
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Effect of metoprolol CR/XL in chronic heart failure: Metoprolol CR/XL Randomised Intervention Trial in Congestive Heart Failure (MERIT-HF). Lancet. 1999 Jun 12;353(9169):2001-7. PMID 10376614
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II): a randomised trial. Lancet. 1999 Jan 2;353(9146):9-13. PMID 10023943
- [Background] van Veldhuisen DJ, Cohen-Solal A, Bohm M, Anker SD, Babalis D, Roughton M, Coats AJ, Poole-Wilson PA, Flather MD; SENIORS Investigators. Beta-blockade with nebivolol in elderly heart failure patients with impaired and preserved left ventricular ejection fraction: Data From SENIORS (Study of Effects of Nebivolol Intervention on Outcomes and Rehospitalization in Seniors With Heart Failure). J Am Coll Cardiol. 2009 Jun 9;53(23):2150-8. doi: 10.1016/j.jacc.2009.02.046. PMID 19497441
- [Background] Petersson M, Friberg P, Eisenhofer G, Lambert G, Rundqvist B. Long-term outcome in relation to renal sympathetic activity in patients with chronic heart failure. Eur Heart J. 2005 May;26(9):906-13. doi: 10.1093/eurheartj/ehi184. Epub 2005 Mar 10. PMID 15764611
- [Background] DiBona GF, Kopp UC. Neural control of renal function. Physiol Rev. 1997 Jan;77(1):75-197. doi: 10.1152/physrev.1997.77.1.75. PMID 9016301
- [Background] Clayton SC, Haack KK, Zucker IH. Renal denervation modulates angiotensin receptor expression in the renal cortex of rabbits with chronic heart failure. Am J Physiol Renal Physiol. 2011 Jan;300(1):F31-9. doi: 10.1152/ajprenal.00088.2010. Epub 2010 Oct 20. PMID 20962112
- [Background] SMITHWICK RH. Hypertensive vascular disease; results of and indications for splanchnicectomy. J Chronic Dis. 1955 May;1(5):477-96. doi: 10.1016/0021-9681(55)90061-8. No abstract available. PMID 14367447
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036